CLINICAL TRIAL: NCT01512940
Title: Laparoscopic Greater Curvature Plication for Weight Loss and Resolution of Diabetes and Other Comorbidities.
Brief Title: Resolution of Comorbidities, Safety and Efficacy of Greater Curvature Plication in Obese Patients.
Acronym: LGCP
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Singh, Kuldeep, M.D., P.A. (Individual)
Responsible Party: Principal Investigator, Kuldeep Singh, Principal Investigator, Singh, Kuldeep, M.D., P.A.
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RPN 2011-024
Record Dates: First submitted 2012-01-15; First posted 2012-01-19 (Estimated); Last update posted 2012-03-13 (Estimated); Status verified 2012-03

CONDITIONS: Obesity
Keywords: obesity; Laparoscopic Greater Curvature Plication; Percent Excess weight Loss; comorbidities; BMI; Bariatric Surgery
MeSH Terms: conditions — Obesity | interventions — Bariatric Surgery

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Procedure: Laparoscopic Greater Curvature Plication — The greater curvature of the stomach is separated from the greater omentum. At least two rows of at least five continuous stitches will be placed about the greater curvature of the stomach starting at or near the angle of His and ending in the antrum. An endoscope will be used to maintain a lumen during the procedure. The two tissue bites of an individual stitch will be centered about the intended fold line.
  Subsequent stitches will be uniformly spaced distally along the length of the fold. The second row of sutures will be placed across the fold line created by the previous row of sutures in the same fashion as the first row. Up to 2 additional rows may be added as required to achieve this result (for a total of up to 4 rows). Upon completion of the procedure, the section of the stomach infolded by the sutures will be inspected using the endoscope.
  Other Names: Bariatric Surgery

SUMMARY:
Various gastric restrictive procedures have evolved over the years but abandoned due to poor long term weight loss, food intolerance or severe gastroesophageal reflux. Laparoscopic gastric plication or laparoscopic greater curvature placation ( LGCP) has recently been done as an alternative to the other restrictive procedures. But the short and long term safety and efficacy outcomes of LGCP is not well documented in current literature. American society of metabolic and bariatric surgery ( ASMBS) guidelines state that LGCP procedures should be considered investigational at this time and should be performed under a study protocol with third party oversight (e.g. IRB) to ensure continuous evaluation of patient safety and to review adverse events and outcomes.

The objective of this study will be to demonstrate feasibility , short term and long term safety and efficacy of LGCP . This will be done by achieving gastric restriction by infolding of stomach and thereby achieving good weight loss .

DETAILED DESCRIPTION:
Since the acceptance of surgical procedures to achieve a sustainable weight loss, many different procedures has been tried with variable success. Among them , various gastric restrictive procedures have evolved over the years but abandoned due to poor long term weight loss, food intolerance or severe gastroesophageal reflux. Currently, laparoscopic adjustable gastric band ( LAGB) and sleeve gastrectomy are being used with variable acceptance and success. Laparoscopic gastric plication or laparoscopic greater curvature plication ( LGCP) has recently been done as an alternative to the other restrictive procedures. But the short and long term safety and efficacy outcomes of LGCP is not well documented in current literature. American society of metabolic and bariatric surgery ( ASMBS) guidelines state that LGCP procedures should be considered investigational at this time and should be performed under a study protocol with third party oversight (e.g. IRB) to ensure continuous evaluation of patient safety and to review adverse events and outcomes.

A prospective nonrandomized study at Cleveland clinic suggested that a reduction in gastric capacity can be achieved by way of plication of stomach and thereby achieving encouraging weight loss. We intend to study this procedure as an alternative to LAGB or sleeve gastrectomy for carefully selected patients. The objective of this study will be to demonstrate feasibility , short term and long term safety and efficacy of LGCP . This will be done by achieving gastric restriction by infolding of stomach and thereby achieving good weight loss . The subjects will be followed up post operatively to observe the effect on the comorbidities along with sustained weight loss. The inclusion and exclusion criteria , target population, duration of subject participation and primary endpoints will be defined and all the data will be recorded per protocol.

ELIGIBILITY:
Inclusion Criteria:

1. Subject is willing to give consent and comply with evaluation and treatment schedule;
2. 18 to 65 years of age (inclusive);
3. Have a BMI > 27 with one or more significant co-morbid medical conditions which are generally expected to be improved, reversed, or resolved by weight loss. These conditions may include but are not be limited to -

   * Hyperlipidemia
   * Type 2 diabetes
   * Mild obstructive sleep apnea
   * Hypertension
   * Osteoarthritis of the hip or knee
4. Agree to refrain from any type of weight-loss drug (prescription or OTC) or elective procedure that would affect body weight for the duration of the trial;
5. HbA1C < 11%
6. For subjects who have Type 2 diabetes, the anti-diabetic medication regimen is no more complex than oral metformin plus one oral sulfonylurea plus once daily insulin injection.
7. Ability to self pay for the procedure and follow up.

Exclusion Criteria:

1. Previous malabsorptive or restrictive procedures performed for the treatment of obesity;
2. Scheduled concurrent surgical procedure, with the exception of SOC liver biopsy;
3. Women of childbearing potential who are pregnant or lactating at the time of screening or at the time of surgery;
4. Any condition which precludes compliance with the study;
5. History or presence of pre-existing autoimmune connective tissue disease
6. Use of prescription or over the counter weight reduction medications or supplements within thirty days of the Screening Visit or the duration of study participation.
7. Psychiatric disorders that may affect compliance with the clinical trial, including dementia, active psychosis, severe depression requiring > 2 medications, or history of suicide attempts. Any condition which places the subject at undue risk for the procedure (surgeon's discretion).

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2011-10; Primary Completion 2012-10 (Estimated); Study Completion 2014-10 (Estimated)

PRIMARY OUTCOMES:
Percent excess weight loss | 3 years
  The percent excess weight loss at 3-years from the time of surgery. The primary analysis will include all available data at the 3-year follow-up.

SECONDARY OUTCOMES:
Resolution of comorbidities | 3 years
  The following comorbidities will be assessed at regular intervals: diabetes, dyslipidemia, liver dysfunction, and hypertension. Measures will include glycosylated hemoglobin, triglycerides, low-density lipoprotein, high-density lipoprotein, serum albumin, liver transaminases, systolic and diastolic blood pressures.

CONTACTS AND LOCATIONS:
Overall Officials: Kuldeep Singh, MD, Principal Investigator — Kuldeep Singh, MDPA
Locations (1):
- Saint Agnes Hospital, Baltimore, Maryland, United States